CLINICAL TRIAL: NCT06021028
Title: Performance of GIOMER Based Resin Composite Restorations Versus Conventional Nanohybrid Resin Composite Restorations in Complex Proximal Carious Cavities in Posterior Teeth. (A 24-month Randomized Clinical Trial)
Brief Title: Performance of GIOMER Based Resin Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, Lecturer, Conservative dentistry department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cons2023
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Controlled Trial. Trial type: Two, Parallel arm design. Trial framework: Equivalence frame Allocation ratio: 1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Triple (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beautifil II Resin composite (Experimental): Giomer restorative
  Interventions: Procedure: complex proximal carious cavities in posterior teeth.
- Neo Spectra resin composite (Active Comparator): Nano-hybrid resin composite
  Interventions: Procedure: complex proximal carious cavities in posterior teeth.

INTERVENTIONS:
Procedure: complex proximal carious cavities in posterior teeth. — Selective enamel etching with 37% phosphoric acid for 30 second will be done then the bonding agent will be applied following the manufacturer's instructions.

SUMMARY:
The aim of the study is to clinically evaluate the performance of GIOMER based resin composite restorations versus conventional nanohybrid resin composite restorations in complex proximal carious cavities in posterior teeth over 2 years follow up. The null hypothesis will be proposed that there will be no difference in the clinical performance of GIOMER based resin composite restorations versus conventional nanohybrid resin composite restorations in complex proximal carious cavities in posterior teeth over 2 years follow up.

DETAILED DESCRIPTION:
Scientific background:

One of the advancements in resin composite technology to support its use as a bioactive material, is the evolution of GIOMER based resin composite material which has an added benefit of sustained fluoride and other ions release and rechargeability. A distinguishing feature of the "giomer" class of restorative materials is the stable surface prereacted glass core (sPRG) that is lined with an ionomer in a resin matrix. This configuration enables the glass core to be protected from moisture, giving it long term aesthetics and the durability of conventional resin composites with ion release and recharge1. When evaluating the clinical performance of low shrinkage giomer based resin composite (Beautifil II LS; Shofu Inc.) compared with a conventional nanohybrid resin composite in class I and class II cavities, It was found that in both groups, according to FDI criteria, the restorations were mostly rated with best scores (Score 1 or 2) regarding the biological, functional, and optical parameters 2. Also, after five years of clinical performance, both the nano-hybrid giomer restorative materials flowable giomer (Beautifil Flow Plus F00; Shofu Inc.) and the conventional nano-hybrid giomer restorative material (Beautifil II; Shofu Inc.) were comparably acceptable and not significantly different for any of the parameters evaluated in occlusal cavities 3. Meanwhile in a recent systematic review, it was concluded that GIOMER based resin composites showed similar clinical performance concerning marginal adaptation and better surface roughness when compared to Resin-modified glass ionomer cement 4.

Statement of the problem:

The survival rate for resin-based composite restorations declined to roughly 85-90% after ten years. Bulk fractures and wear, which accounted for about 70% of replacements, were the main causes of restorative replacement. About 20% of the resin-based restorations were replaced because of caries at the margins of the restorations, and 10% were due to retention loss, poor color matching, poor marginal integrity, endodontic therapy, or cusp fracture 5. These failures are correlated mainly with patient risk profile i.e., caries risk , presence of parafunctional habits and those with high number of restored surfaces (complex cavities) 6.

Rationale:

In a retrospective study7, the percentage of clinically satisfactory complex Class II resin composite was 78% after five years. The main reasons for the failure presented were related to the fracture of the restoration (Bravo-16%) and defective marginal adaptation (Charlie-8.2%). Although many studies have evaluated the clinical performance of GIOMER based resin composite 2-4, none of them evaluated its clinical performance in complex Class II cavities, up till now, where the restorations are subjected to high stress conditions.

External validity:

Offering the patient, a bioactive giomer based restoration with an added benefit of sustained remineralizing fluoride and other ions release also rechargeability while on the same time it has the long term aesthetics and clinical longevity of conventional resin composite restorations.

Choice of the comparator:

A conventional nanohybrid resin composite material will be used as the comparator as it gives an accepted long term clinical performance according to a recent systematic review 7. Aim of the study:

The aim of the study is to clinically evaluate the performance of GIOMER based resin composite restorations versus conventional nanohybrid resin composite restorations in complex proximal carious cavities in posterior teeth over 2 years follow up.

Methods:

Study Settings:

This clinical trial will be held in Conservative dentistry department clinic, Faculty of Dentistry- Cairo University, Egypt.

Sample size Calculation:

The sample size was calculated based on a previous study by Torres et al in 2020, in which percentage of clinically excellent large class 2 restorations regarding fracture and retention was 87.5%. By implementing a two tailed Z test for difference between two independent proportions with an alpha level of 5% and a power of 80%. The minimum sample size needed was 34 per group in order to detect a difference of 30%. Sample size was increased by 10% to compensate for possible dropouts to reach 38 teeth per group. Sample size was performed using G*Power version 3.1.9.2 for windows.

Methods: Assignment of interventions

Allocation:

Sequence generation:

Simple randomization will be made by a contributor, who will not be further involved in any of the phases of the clinical trial, to generate random numbers using Random Sequence Generator, Randomness and Integrity Services Ltd (https://www.random.org/).

Allocation concealment:

The operator will choose between random numbers placed in an opaque sealed envelope.

Blinding:

The participants and both assessors will be blinded to the type of the material used and the application technique.

Interventions:

After profound local anesthesia, conservative cavity preparations will be performed with highspeed burs under constant cooling. The cavity outline and carious tissue will be removed following the recent conservative cavity preparation and caries excavation guidelines. All restored teeth will be isolated using a rubber dam. After applying the suitable matrix system and wooden wedge.

Intervention group:

Selective enamel etching with 37% phosphoric acid for 30 second will be done then the bonding agent (BeautiBond Universal, Shofu, Inc., Japan) will be applied following the manufacturer's instructions. The restorative material (Beautifil II, Shofu, Inc., Japan ) will be inserted into the cavity which is converted into a class I configuration using a centripetal build-up sequence and light cured following the manufacturer's instructions, then finished and polished after occlusion adjustment.

Comparator group:

The universal bonding agent ( Prime and Bond Active, Dentsply Sirona ) will be applied following the manufacturer's instructions with previous selective enamel etching with 37% phosphoric acid for 30 seconds. The restorative material (Neo Spectra, Dentsply Sirona) will be inserted into the cavity as mentioned before and light cured following the manufacturer's instructions, then finished and polished after occlusion adjustment.

Data collection methods:

*Baseline data collection: For every patient medical and dental history will be obtained. All patients will be given oral hygiene instructions before operative treatment, and they will be referred to the periodontology department for scaling and polishing prior restorative procedures if needed.

*Outcome data collection: FDI criteria for clinical evaluation of dental restoration will be used by the two assessors. If they differ in the evaluation score, they will discuss together till reaching a consensus.

Patient retention:

The patients' phone number will be recorded in their charts. Before the follow up visit, the patient will receive a reminder phone call by If the patient did not answer, another appointment will be scheduled within a week.

Data management:

All data of the trial will be stored on a computer and encrypted using a password. Data will be backed up on cloud storage to prevent it from being lost.

Statistical methods:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 25 (SPSS Inc., Chicago, IL). Numerical data will be represented as mean and standard deviation or median and range. Categorical data will be represented as numbers and percentages. Data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the Student's t-test while for non normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. An equivalence limit will be tested. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Harms:

The operator would inform the participants about any possible harm (post-operative hypersensitivity or fracture of the restoration). If present, participants are instructed to contact the operator immediately by a phone call.

Research ethics approval Application forms for conducting clinical trials, checklist and informed consent of the Research Ethics Committee (REC) Faculty of Dentistry, Cairo University will be fulfilled, this is to prevent any unethical management or harms during the study toward the participants. The operator will be responsible for obtaining the informed consents from the participants during the enrollment day.

Protocol amendments If a new protocol will be used a protocol amendment will be registered with a copy of the new protocol and an explanation about the reasons for it. If there is a change in this protocol that affects trial ethics or the scientific content of the trial, an amendment with brief explanation will be also submitted.

Confidentiality The personal data of the participants will not present on the protocol form and it would be secured for 10 years after the trial to protect their privacy.

Declaration of interests There is no conflict of interest. Funding is accepted from Shofu, Inc., Japan and Ivoclar Vivadent, Schaan, Liechtenstein.

Ancillary and post-trial care Patients will be followed up after the restorative work to maintain the oral hygiene measures. When there is any evidence of restoration failure, patients will be treated by immediate restoration replacement by different restorative option to the tooth.

Dissemination policy Full protocol will be published online in www.clinicaltrials.gov to keep the integrity of the research methods and to avoid repetition. The results of this clinical trial will be internationally published.

Declaration of originality:

This research has not been submitted to any other universities, institutions or even persons for the award of any degree, diploma, or publication any time before.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria of participants:

1. Patients with proximal carious cavities in molars.
2. 18 - 50 years.
3. Males or Females.
4. Good oral hygiene.
5. Co-operative patients approving to participate in the study.

Inclusion Criteria of teeth:

1. Pulp asymptomatic vital carious complex class II upper or lower posterior teeth.
2. The presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

   -

   Exclusion Criteria:
   * Exclusion criteria of participants:

   Poor oral hygiene. Severe medical complications. Pregnancy. Allergic history concerning methacrylates Heavy smoking. Xerostomia. Lack of compliance. Evidence of parafunctional habits Temporomandibular joint disorders.

   Exclusion criteria of the teeth:

   Teeth involving more than three surfaces and indicated for indirect restorations.

   Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis. Severe periodontal problems.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Fracture & retention | 24 months
  FDI criteria Functional properties

SECONDARY OUTCOMES:
Rest of FDI criteria | 24 months
  FDI criteria Functional properties

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Hesham Abd ElAziz, Phd, Principal Investigator — Cairo University
Locations (1):
- Mohamed Mohamed sabry Mohamed, Cairo, Nasr City, Egypt